CLINICAL TRIAL: NCT01608555
Title: Tobramycin 300 mg o.d. Aerosol in in Adult Patients With Cystic Fibrosis: Pilot Study on Antimicrobial Activity
Brief Title: Tobramycin 300 mg Once-a-day (o.d.) Aerosol in Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Francesco Blasi, Professor of respiratory medicine, University of Milan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP2; 2011-001821-26 (EudraCT Number)
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; bacterial load; inhaled tobramycin
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- inhaled tobramycin once-a-day (Experimental): Adult patients, with cystic fibrosis, requiring inhaled tobramycin prophylaxis. Patient will be treated with a single dose of 300 mg tobramycin od for 28 days.
  Interventions: Drug: tobramycin

INTERVENTIONS:
Drug: tobramycin — inhaled tobramycin 300 mg single dose OD for 28 days
  Other Names: Bramitob

SUMMARY:
The study will include 10 adult patients with cystic fibrosis. The aim of the study is to evaluate whether Tobramycin 300 mg aerosol once-a-day for 28 days can reduce the bacterial load in the airways. Secondary end-point is the evaluation of variation in bacterial susceptibility during and at the end of study period.

DETAILED DESCRIPTION:
Ten adult patients with cystic fibrosis will be enrolled in a stable phase and will received prophylaxis with aerosol of Tobramycin 300 mg once a day for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, male and female, age range 18-45 years
* Diagnosis of cystic fibrosis
* FEV1 >50% predicted.
* sputum samples available
* Chest x ray negative for pneumonia and tuberculosis
* Informed consent

Exclusion Criteria:

* Allergy to tobramycin
* Use of systemic steroids in the previous 2 weeks
* Pregnancy or breast feeding
* Treatment with other experimental drug in the previous 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of bacterial load decrease | day 7-9 vs day 1, day 14-16 vs day 7-9, day 28-30 vs day 14-26
  Bacterial load in sputum will be evaluated during and at the end of treatment

SECONDARY OUTCOMES:
Evaluation of inflammatory serum biomarker | day7-9 vs day 1, Day 14-16 vs day 7-9, Day 28-30 vs 14-16
  Serum levels of biomarker (PCT) will be evaluated during and at the end of treatment
Evaluation of serum biomarker | day7-9 vs day 1, Day 14-16 vs day 7-9, Day 28-30 vs 14-16
  Evaluation of C-reactive protein levels during and at the end of treatment
Evaluation of serum biomarker | day7-9 vs day 1, Day 14-16 vs day 7-9, Day 28-30 vs 14-16
  Evaluation of KL6 levels during and at the end of treatment
evaluation of serum biomarker | day7-9 vs day 1, Day 14-16 vs day 7-9, Day 28-30 vs 14-16
  Evaluation of interleukin 6 during and at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Pizzamiglio, MD, Principal Investigator — University of Milan Italy
Locations (1):
- IRCCS Ospedale Maggiore Policlinico via F. Sforza 35, Milan, Italy